CLINICAL TRIAL: NCT05406778
Title: SPARK Neuro Quantitative Resting State EEG Protocol for Assessing Cognitive Impairment and Alzheimer's Disease Status- The REMIND Study
Brief Title: The REMIND Study- SPARK Neuro Software Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Neuro Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1001
Record Dates: First submitted 2022-05-26; First posted 2022-06-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Cognitive Impairment
Keywords: EEG; Electroencephalography; Machine learning
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Subjects - Variable Cognitive Status (Other): Subjects meeting Inclusion/Exclusion criteria with open eyes/closed eyes EEG collection.
  Interventions: Device: SPARK Test

INTERVENTIONS:
Device: SPARK Test — Thirty (30) minutes of resting state EEG data collection.

SUMMARY:
The study utilizes investigational software, the SPARK Test, with an FDA-cleared electroencephalography (EEG) amplifier and EEG cap to collect and patient EEG data.

DETAILED DESCRIPTION:
The aim of this study is to collect data to support development of an algorithm to determine whether applying machine-learning techniques to eyes open/eyes closed resting-state electroencephalography (EEG) can characterize patient's cognitive status and detect the presence or absence of AD on the basis of the patient's EEG.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 to 85 at the time of consent
2. Informant available and willing (remotely or in-person) to provide information about sleep patterns and cognitive functioning who spends >8 hours per week with primary subject
3. Subject or Legally Authorized Representative (LAR) has the ability to provide informed consent and comply with the protocol.

Exclusion Criteria:

1. Unable to remain still for up to 30 minutes during EEG data recording
2. Subjects currently on and unable to wash out concomitant medications, including: 1) opiates; 2) benzodiazepines and nonbenzodiazepine hypnotics; 3) sedative antihistamines; 4) tricyclic anti-depressants; 5) skeletal muscle relaxants; 6) antiepileptics; 7) antipsychotics; 8) antimanic agents; 9) THC; 10) anticholinergics
3. Previous history of craniotomy
4. Medical or psychiatric illness that would interfere with study participation
5. History of epilepsy or chronic seizure disorder
6. Presence of non-dental metal in head
7. Currently experiencing a skin disease on scalp that would affect electrode contacts
8. Subject meets at least one of the following criteria:

   1. Diagnosis of cognitive impairment from various underlying pathologies as indicated by one of the diagnostic codes listed in Appendix A (protocol)
   2. MMSE score of 27 or less
   3. Treating physician or PI have documented that the patient is cognitively impaired, with judgment of cognitive impairment having been made within the 6 months prior to enrollment
9. Substance Use Disorder, including Alcohol

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
EEG Data collection for AI software development | During the diagnostic procedure
  Rate of complete software collection per enrolled subjects complete a SPARK Test recording.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Island Psych, Loma Linda, California
  - CenExel Rocky Mountain, Englewood, Colorado
  - Renstar Medical, Ocala, Florida
  - Arcturus Healthcare PLC, Troy - Internal Medicine Division, Troy, Michigan
  - Alivation Health, Lincoln, Nebraska
  - Advanced Neuro, El Paso, Texas
  - Integrated Neurology, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No